CLINICAL TRIAL: NCT03966742
Title: Doxorubicin Eluting Intra-arterial Embolization for Aggressive Desmoid Fibromatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Eldad Elnekave, MD, Director, Clinic Interventional Oncology, Rabin Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC-0485-17
Record Dates: First submitted 2019-04-08; First posted 2019-05-29 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Desmoid; Desmoid Fibromatosis of Skin; Desmoid Neoplasm of Chest Wall; Desmoid Tumor Caused by Somatic Mutation; Aggressive Fibromatoses; Fibromatosis Desmoid; Desmoid Fibromatosis
MeSH Terms: conditions — Desmoid Tumors; Desmoid disease, hereditary

STUDY DESIGN:
Intervention Model Description: All patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Doxorubin-eluting particle embolization for treatment of Desmoid Fibromatosis.
  Interventions: Procedure: Drug Eluting Bead Embolization (DEB) for Desmoid Fibromatosis

INTERVENTIONS:
Procedure: Drug Eluting Bead Embolization (DEB) for Desmoid Fibromatosis — Delivery of Doxorubicin selectively into Desmoid Fibromatosis utilizing its vascular supply as a conduit, and ionic loading the doxorubicin onto embolized particles as the drug delivery vehicle.
  Maximal dose is 75 mg/m2 and at least 50 mg. The bead size is 75-300 Mµ in a 2 CC syringe.

SUMMARY:
In this study Drug-eluting microbeads (DEB) loaded with Doxorubicin will be delivered into the target Desmoid Fibromatoses (DF) tissue via selective arterial embolization by angiographic technique. The objective of the study is to demonstrate the safety and efficacy of this treatment.

DETAILED DESCRIPTION:
Desmoid Fibromatoses (DF) are locally aggressive lesions associated with substantial morbidity and potentially mortality, due to invasion of adjacent neurovascular structures and vital organs. They have no potential for metastasis. Histologically, they are characterised by mature fibroblasts within a matrix of abundant fibrous stroma. While 5-15% of cases are seen in patients with Familial Adenomatous Polyposis (FAP) syndrome, the vast majority arise sporadically.

The etiology of Desmoids remains poorly understood and the therapeutic approaches in their management remain very diverse. For resectable lesions, surgery is recommended but reported cure rates range broadly from 12-80%. Systemic treatments range from non-steroidal anti-inflammatories and anti-estrogenic therapy to targeted tyrosine kinase inhibitors and cytotoxic chemotherapy, most commonly methotrexate, vinblastine and doxorubicin.

Doxorubicin is an anthracycline with demonstrated efficacy in treating desmoids at systemic IV doses of 50- 75mg/m2 over 3-4 week cycles. Extended use is limited by dose - dependent cardiotoxicity which can be seen in up to 36% of patients receiving doses in excess of 550mg/m2. Delayed cardiotoxicity is particularly common and less predictable among pediatric cancer survivors.

Selective trans-arterial chemo-embolization (TACE) is a method to achieve high tissue drug concentration with minimal systemic toxicity. Historically, this has been achieved by mixing doxorubicin with embolic agents such as lipiodol or gelatin sponge in the treatment of hepatocellular carcinoma (HCC).

Drug-eluting microbeads (DEB) ionically loaded with doxorubicin have shown sustained release in TACE target tissues with substantially lower serum drug concentrations when compared to lipiodol TACE.

The present study utilizes DEB's loaded with Doxorubicin delivered into the target DF tissue via selective arterial embolization by angiographic technique. This study follows a successful feasibility study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-80 years.
2. Histologically confirmed diagnosis of Desmoids Fibromatosis.
3. After at least one systemic treatment line. Standard first line systemic treatment may include: Methotrexate, Vinblastine, Doxorubicin, Liposomal Doxorubicin (Doxil), NSAIDS or hormonal treatment. If first line treatment is renounced, this treatment decision must be documented. Considering the trend of avoiding surgical treatment, the documentation must include that the treatment decision is not associated to the resectability of the tumor.
4. Karnofsky performance status (PS)>50% for patients older than 16 years or Lansky PS >50% for patients under 16 years.
5. At least one measurable lesion, with a long diameter of at least 30mm, with an anatomical location accessible for endovascular treatment.
6. T2 signal increase on MRI.
7. No evidence of prior treatment toxicity, adequate washout period after prior treatment:

   * 14 days after myelosuppressive chemotherapy treatment.
   * 7 days after GCSF (Granulocyte colony-stimulating factor), 14 days after Neulastim.
   * 7 days after targeted/biologic treatment.
8. Female patients of childbearing potential must be willing to use an adequate method of contraception (hormonal, barrier or abstinence) for the treatment period and up to 90 days after the treatment completion.
9. Willing and able to provide written informed consent for the trial.

Exclusion Criteria:

1. Participation in another interventional study.
2. Congestive heart failure, characterised by LVEF (Left Ventricular Ejection Fraction) < 50% or Shortening fracture < 27%.
3. Previous treatment with anthracycline of a accumulative dose of more than 360 mg/m2.
4. History of allergic reaction attributed to Doxil or doxorubicin treatment.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness, social situations that would limit compliance with study requirements.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Objective response rate of tumor size. | At baseline ; 6-10 weeks after each treatment
  Response to treatment. Measured by change in tumor size according to RECIST (Response Evaluation Criteria in Solid Tumors) version 1.1 criteria.
Objective response rate of tumor biological activity. | At baseline ; 6-10 weeks after each treatment
  Response to treatment. Tumor biological activity measured by change in MRI T2 signal intensity.
Patient reported outcomes. | At baseline ; 6-10 weeks after each treatment
  Change in clinical symptoms measured by standard clinical patient questionnaires - EORTC QLQ-C30. (Quality of Life Questionnaire).
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high level of functioning, a high score for the global health status / QoL represents a high QoL. Similarly, a high score for a symptom scale represents a high level of symptomatology.

SECONDARY OUTCOMES:
Adverse event profile (safety) | At baseline ; 6-10 weeks
  Treatment safety measured by standard patient questionnaires and clinical evaluation using CTCAE (Common Terminology Criteria for Adverse Events) version 5.0.

OTHER OUTCOMES:
Pharmacokinetics of Doxorubicin | 5 minutes, 30 minutes, 1 hour, 12 hours, 24 hours after treatment procedure
  Measurements of blood Doxorubicin concentration (mg/ml) over time, after treatment.
Exploratory biomarkers | At baseline ; 6-10 weeks
  Immunohistochemistry assay assessing the staining pattern (marked as negative to mildly or strongly positive) for: beta-catenin, keratin, SMA (smooth muscle actin). Ki-67 staining will be scored by percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elnekave E, Atar E, Amar S, Bruckheimer E, Knizhnik M, Yaniv I, Dujovny T, Feinmesser M, Ash S. Doxorubicin-Eluting Intra-Arterial Therapy for Pediatric Extra-Abdominal Desmoid Fibromatoses: A Promising Approach for a Perplexing Disease. J Vasc Interv Radiol. 2018 Oct;29(10):1376-1382. doi: 10.1016/j.jvir.2018.04.009. Epub 2018 Jul 31. PMID 30075974